CLINICAL TRIAL: NCT06586177
Title: Understanding the 'Durable Effect' Concept of B-cell Modulating Therapies
Acronym: REBELLION-MS
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Dr rer. nat. Sven Meuth, Chairman, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2021-1475
Record Dates: First submitted 2024-07-04; First posted 2024-09-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 (C1; basic cohort): Participants will be seen every 6 months up until month 24, then every 12 months. The following parameters will be collected: demographic data, disease characteristics incl. EDSS and MRI data, serum samples, and PBMCs. Furthermore, SF-36 and FSMC are documented.
  Interventions: Drug: Anti-CD20 antibody
- Cohort 2 (C2; in-depth cohort): In addition to the parameters collected for C1, participants of C2 will receive: clinical evaluation incl. EDSS and sampling of serum and PBMCs at months 1 and 3, MFSC every 6 months, and OCT as well as NPT every 12 months.
  Interventions: Drug: Anti-CD20 antibody

INTERVENTIONS:
Drug: Anti-CD20 antibody — Study participants receive an anti-CD20 antibody according to the summary of product characteristics.

SUMMARY:
This prospective, observational clinical study aims to longitudinally assess peripheral immune cell profiles of patients with relapsing-remitting multiple sclerosis (RRMS) receiving anti-CD20 therapy with ofatumumab (OFA), ocrelizumab (OCR), ublituximab (UBX), and rituximab (RTX). Throughout the study, clinical data - including relapse events, patient scores, and neuropsychological parameters - will be collected, along with results from imaging techniques such as Optical Coherence Tomography (OCT) and Magnetic Resonance Imaging (MRI). This clinical data will be combined with immunological analyses, including multidimensional flow cytometry (mFC), bulk RNA sequencing (bulk-Seq), T and B cell receptor sequencing (TCR/BCR-Seq), proteomics, and immunoglobulin analysis. This approach aims to enable a detailed characterization of changes in the immune cell repertoire and their impact on the clinical disease course.

DETAILED DESCRIPTION:
B cell targeted therapies have become a key element in the treatment of multiple sclerosis due to their effectiveness in rapid and long-lasting depletion of B cells in peripheral blood (PB), significantly reducing relapse rates and disability progression. The monoclonal antibodies OFA, OCR, UBX, and RTX target the B cell surface protein CD20, however it is unclear how B cell depletion and subsequent repopulation allows for immune system reconstitution and how other immune cell populations are affected by these therapies. Furthermore, the relevance of immune cell changes - beyond B cell depletion - for clinical disease stability remains insufficiently understood.

By collecting comprehensive and structured prospective clinical data alongside immunological analyses, this study aims for a better understanding of immunological changes in RRMS patients receiving anti-CD20 therapies and the implications of those alterations in immune cell profiles on the clinical disease course. REBELLION-MS plans for two patient cohorts: cohort 1 (C1; basic cohort) and cohort 2 (C2; in-depth cohort). Participants in C1 will be seen every 6 months up until month 24, then every 12 months. The following parameters will be collected: demographic data, disease characteristics incl. Expanded Disability Status Scale (EDSS) and magnetic resonance imaging (MRI) data, serum samples, and Peripheral Blood Mononuclear Cells (PBMCs). Furthermore, Short Form-36 (SF-36) and Fatigue Scale for Motor and Cognitive Functions (FSMC) are documented. Participants of C2 will receive additional evaluations: clinical evaluation incl. EDSS and sampling of serum and PBMCs at months 1 and 3, Multiple sclerosis functional composite (MFSC) every 6 months, and optical coherence tomography (OCT) as well as neuropsychological assessment (NPT) every 12 months. Serum samples and PBMCs will be analyzed by mFC, bulk-Seq, TCR/BCR-Seq, and proteomics, among other methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed relapsing-remitting multiple sclerosis (RRMS) according to 2017 revised McDonald criteria
* Current treatment with B cell modulating therapies or initiation/transition to B cell modulating therapies according to the "Summary of Product Characteristics (SmPC)"
* EDSS score of 0.0 to 7.0

Exclusion Criteria:

* Previous treatment with alemtuzumab, cladribine, cyclophosphamide, mitoxantrone, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, total body irradiation or bone marrow transplantation
* Medical, psychiatric, cognitive, or other conditions that, in the opinion of the investigator, impair the patient's ability to understand the patient information and give informed consent
* Patients receiving immunosuppressive treatment for conditions other than MS or long-term corticosteroid treatment
* Patients with confirmed infection by the Human Immunodeficiency Virus or Hepatitis C Virus

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The study population will include RRMS patients receiving B cell modulating therapies.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the peripheral immune cell profile | Baseline up to 48 months
  Immune cell subpopulations will be analyzed longitudinally by multidimensional flow cytometry [% of all living cells and mean fluorescent intensity of different cell surface markers].
Change from baseline in protein profile of the peripheral blood | Baseline up to 48 months
  Protein expression will be measured longitudinally using proteomics.
Change from baseline in TCR/BCR profile | Baseline up to 48 months
  T cell and B cell receptor profile will be measured longitudinally using BCR- and TCR-sequencing.

SECONDARY OUTCOMES:
Change from baseline in Expanded Disability Status Scale (EDSS) Score | Baseline up to 48 months
  The EDSS is used to quantify disability due to symptoms of MS and to track changes in disability status over time. Scores range from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). Higher scores indicate a greater level of disability.
Change from baseline in Short Form Health Survey (SF-36) | Baseline up to 48 months
  The SF-36 questionnaire is used to measure health-related quality of life summarized into two overarching scales: physical health and mental health. It contains 36 questions including eight subscales that capture various aspects of health and well-being. For each of these subscales, multiple questions are asked, each rated on a scale from 0 to 100, with higher scores indicating better health and higher levels of well-being.
Change from baseline on Magnetic Resonance Imaging (MRI) | Baseline up to 48 months
  Cerebral MRI (cMRI) and spinal MRI (sMRI) performed as part of the clinical routine workup will be analyzed and quantified for the number of lesions, new lesions, and active lesions.
Change from baseline in Retinal Nerve Fiber Layer thickness (RNFL) | Baseline up to 48 months
  Retinal Nerve Fiber Layer thickness (RNFL) will be measured longitudinally by Optical Coherence Tomography (OCT).
Change from baseline in visual acuity (HCV and LCV) | Baseline up to 48 months
  High-contrast visual acuity (HCV) and low-contrast visual acuity (LCV) are measured longitudinally in both eyes.
Change from baseline in Fatigue Scale for Motor and Cognitive Functions (FSMC) | Baseline up to 48 months
  Fatigue is rated using the self-administered 20-item FSMC questionnaire that includes ten questions related to motor fatigue and ten questions related to cognitive fatigue. A Likert-type 5-point scale produces a score between 1 and 5 for each scored question. Minimum value is 20 (no fatigue at all) and maximum value is 100 (severe fatigue). Higher scores indicate higher fatigue.
Change from baseline in Multiple Sclerosis Functional Composite (MSFC) Score | Baseline up to 48 months
  MSFC has 3 components: 1. Timed 25-foot walk (T25FW), 2. 9-hole peg test (9HPT) [dominant and nondominant hands], and 3. Paced Auditory Serial Addition Test (PASAT).
  The MSFC Z-score is calculated by creating Z-scores for each component of the MSFC and averaging them to create an overall composite score.
  MSFC Z-score = (Z25-foot-walk + Z9HPT+ ZPASAT)/3. A Z-score represented the number of standard deviations participant's test result was higher (Z > 0) or lower (Z < 0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes.
Change from baseline in Symbol Digit Modalities Test (SDMT) | Baseline up to 48 months
  The Symbol Digit Modalities Test (SDMT) assesses information processing speed and attention. It involves matching symbols to numbers according to a given key within a specified time limit.
  Z-Scores are calculated. A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes.
Change from baseline in Verbal Memory Learning Test (VMLT) | Baseline up to 48 months
  Verbal Memory Learning Test (VMLT) is an examination of verbal learning and memory by presenting a list of words to the participant multiple times and then asking them to recall as many words as possible after each presentation.
  A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes.
Change from baseline in Brief Visuospatial Memory Test (BVMT) | Baseline up to 48 months
  Brief Visuospatial Memory Test (BVMT) assesses visuospatial learning and memory. Participants are asked to recall a series of abstract designs after multiple presentations. A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes.
Change from baseline in Montreal Cognitive Assessment (MoCA) | Baseline up to 48 months
  Montreal Cognitive Assessment (MoCA) ranges from 0 - 30, the higher the number the better the cognitive function.
Change from baseline in BDI-FS/BDI II | Baseline up to 48 months
  Beck Depressions-Inventar (Fast-Score) (BDI-FS/BDI II) assesses depressive symptoms. Higher scores indicate more severe signs of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich-Heine University, Duesseldorf, Düsseldorf, Germany

REFERENCES:
- [Derived] Willison AG, Hagler R, Weise M, Elben S, Huntemann N, Masanneck L, Pfeuffer S, Lichtenberg S, Golombeck KS, Preuth LM, Rolfes L, Ozturk M, Ruck T, Melzer N, Korsen M, Hauser SL, Hartung HP, Lang PA, Pawlitzki M, Rauber S, Meuth SG. Effects of Anti-CD20 Antibody Therapy on Immune Cell Dynamics in Relapsing-Remitting Multiple Sclerosis. Cells. 2025 Apr 6;14(7):552. doi: 10.3390/cells14070552. PMID 40214505